CLINICAL TRIAL: NCT00233948
Title: A Phase I/II Study of Nelfinavir in Liposarcoma
Brief Title: Nelfinavir Mesylate in Treating Patients With Recurrent, Metastatic, or Unresectable Liposarcoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug availability issues
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04090; NCI-2010-01263; CDR0000438712 (Registry Identifier: PDQ); FDA R01FD003006-03 (Other: FDA Office of Orphan Products Development)
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Adult Liposarcoma; Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Liposarcoma; Sarcoma | interventions — Nelfinavir; Biopsy; Gene Expression Profiling; Blotting, Western; Reverse Transcriptase Polymerase Chain Reaction; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral nelfinavir mesylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: nelfinavir mesylate; Procedure: biopsy; Other: laboratory biomarker analysis; Other: pharmacological study; Genetic: gene expression analysis; Genetic: western blotting; Genetic: reverse transcriptase-polymerase chain reaction; Other: immunoenzyme technique

INTERVENTIONS:
Drug: nelfinavir mesylate — Given orally
  Other Names: Viracept
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Genetic: gene expression analysis — Correlative studies
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques

SUMMARY:
RATIONALE: Antiviral drugs, such as nelfinavir mesylate, may help prevent cancer cells from spreading.

PURPOSE: This phase I/II trial is studying the side effects and best dose of nelfinavir mesylate and to see how well it works in treating patients with recurrent, metastatic, or unresectable liposarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the toxicity and tolerance of nelfinavir in patients with liposarcoma.

II. To define the maximum tolerated dose (MTD) of nelfinavir when given daily as a single agent and to describe the toxicities at each does studied.

III. To evaluate the pharmacokinetics of nelfinavir. IV. To assess the response rate and progression free survival in patients with liposarcoma treated with nelfinavir.

V. To evaluate the expression and activity of certain proteins in the tumors of patients entered on this study, which may be important to the cytotoxicity of nelfinavir (SREBP-1, p21, NFkB (NFkappaB), caspase 3).

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive oral nelfinavir mesylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion

* Patients must have histologically confirmed liposarcoma, which is recurrent, metastatic or unresectable
* There is no limit to prior chemotherapy regimens; in addition, patients may have prior radiation
* All patients must have measurable disease, defined as lesions that can be accurately measured in at least one dimension (>= 20 mm with conventional techniques or >= 10mm with spiral CT scan); pleural effusions and ascites will not be considered measurable, but may be present in addition to the measurable lesion(s)
* ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2; patients should have an expected survival of at least 3 months
* Absolute neutrophil count >= 1,000/ul
* Platelets >= 75000/ul
* Total bilirubin =< 2.0 g/dl
* AST(SGOT)/ALT(SGPT) =< 2.0X institutional upper limit of normal
* Brain metastasis is not an exclusion; however, patients are only eligible if they have had successful control of the brain tumor(s) by surgery or radiation therapy
* All prior therapy must have been completed at least 3 weeks prior to the patient's entry on this trial
* No concurrent chemotherapy, radiotherapy, immunotherapy or other investigational agents
* Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation; should a women become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willingness to sign a written informed consent document

Exclusion

* Patient has had prior treatment with or is currently taking a protease inhibitor
* Patients enrolled cannot be on the following medications: cisapride, triazolam, midazolam, ergot derivatives, amiodarone, quinidine, dihydropyridine calcium antagonists (amlodipine, felodipine, isradipine, nicardipine, nifedipine, nimodipine, and nisoldipine), sildenafil, dilantin, rifampin or oral contraceptives
* Uncontrolled intercurrent illness
* Patients must have recovered from any expected toxicities of previous chemotherapy or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-03; Primary Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Chow, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 1: Oral Nelfinavir at 1250mg bid.
- Phase I: Dose Level II: Oral Nelfinavir at 1500mg bid.
- Phase I: Dose Level III: Oral Nelfinavir at 2125mg bid.
- Phase I: Dose Level IV; Phase II: Oral Nelfinavir at 3000mg bid.
- Phase I: Dose Level V: Oral Nelfinavir at 4250mg bid.
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level II | Phase I: Dose Level III | Phase I: Dose Level IV | Phase I: Dose Level V | Phase II
Started | 4 | 3 | 3 | 3 | 4 | 12
Completed | 3 | 3 | 3 | 3 | 4 | 12
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Phase I dose escalation portion of the study. Initial dose of oral Nelfinavir was 1250 mg bid with escalation to the MTD at 4250 mg bid using a standard 3+3 dose escalation scheme.
- Phase II: Oral Nelfinavir at 3000 mg bid
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 17 | 12 | 29
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 81] | 63 [46 to 84] | 64 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 11 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) (Phase I)
Description: DLT is defined as any grade III toxicity not reversible to grade II or less within one week, or any grade IV toxicity. Hyperlipidemia, hyperglycemia, nausea, vomiting and diarrhea are not DLTs unless they are uncontrolled grade 3/4. Dose delays lasting more than 2 weeks due to toxicity are considered a DLT. Dose escalation schedule for nelfinavir: 1250 mg bid ; 1500 mg bid; 2125 mg bid; 3000 mg bid; 4250 mg bid ; 6000 mg bid ; 8500 mg bid ; 12000 mg bid
Time Frame: 4 weeks from start of treatment, up to 2 years
Population: All patients receiving treatment were evaluated for DLT.
Measure: Number; unit: participants with DLTs
Groups:
- Phase I: Dose Level I: Oral Nelfinavir at 1250mg bid.
Arm/Group | Phase I: Dose Level I | Phase I: Dose Level II | Phase I: Dose Level III | Phase I: Dose Level IV | Phase I: Dose Level V
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4
participants with DLTs | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: The highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. If PK analysis of 3 patients treated at 4250 mg bid and 3 patients at 3000 mg bid confirms that the first dose area under the curve and Cmax of nelfinavir does not increase appreciably at doses greater than 1875 mg BID then 3000 mg BID will be deemed the MTD.
Time Frame: 4 weeks from start of treatment, up to 2 years
Population: All patients observed for 28 days while receiving a full course of therapy or who experienced a DLT. Patients withdrawing before completion of the first course, for reasons other than DLT, were replaced.
Measure: Number; unit: mg
Groups:
- Phase I: All patients enrolled on the Phase I (dose-finding) portion of the study.
Arm/Group | Phase I
Number analyzed (Participants) | 17
mg | 3000

3. Primary Outcome: Overall Response Rate (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: After 3 cycles of treatment, up to 2 years.
Population: Patients who complete 3 cycles of treatment or who terminate treatment for reasons of toxicity, or who progress prior to the completion of 3 cycles of therapy on the Phase II portion of the study.
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 12
participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over a period of 5 years, 2 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Phase I: Dose Level I | Phase I: Dose Level II | Phase I: Dose Level III | Phase I: Dose Level IV | Phase I: Dose Level V | Phase II
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 2/3 | 1/3 | 0/4 | 2/12
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3 | 4/4 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level I (N=4) | Phase I: Dose Level II (N=3) | Phase I: Dose Level III (N=3) | Phase I: Dose Level IV (N=3) | Phase I: Dose Level V (N=4) | Phase II (N=12)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level I (N=4) | Phase I: Dose Level II (N=3) | Phase I: Dose Level III (N=3) | Phase I: Dose Level IV (N=3) | Phase I: Dose Level V (N=4) | Phase II (N=12)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 2 (4) | 1 (1) | 3 (6) | 8 (54)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 7 (8)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 4 (14)
Diarrhea (Gastrointestinal disorders) | 4 (13) | 1 (1) | 3 (6) | 3 (8) | 4 (11) | 10 (48)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (5) | 5 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (8)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 1 (3) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 9 (21)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (9)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 1 (1) | 1 (4) | 3 (10) | 2 (4)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 4 (9) | 5 (11)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 2 (2) | 1 (3) | 3 (7) | 4 (11)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (14)
Hypercholesterolemia (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (8) | 1 (6) | 3 (25)
Leukopenia (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 1 (4) | 1 (3) | 8 (20)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 1 (2) | 2 (13)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (8) | 0 (0) | 4 (10)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (12) | 0 (0) | 1 (4) | 3 (5) | 6 (46)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 8 (17)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (2) | 5 (11)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 2 (5) | 4 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (6)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (8)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 3 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (7)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 7 (18)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 6 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (4)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
After 12 patients were accrued to the Phase II portion, the study was terminated…protocol objectives for the Phase II portion not met. Closed prematurely due to drug availability issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes